CLINICAL TRIAL: NCT04548518
Title: A Phase III Double Blinded, Randomized, Controlled, Non-inferiority Trial to Evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine, in Healthy Thai Subjects Aged 65 Years and Above
Brief Title: Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine, in Healthy Thai Elderly
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Tri Fluvac Vaccine in Elderly
Record Dates: First submitted 2020-08-17; First posted 2020-09-14 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Influenza
Keywords: Influenza Vaccine; Tri Fluvac vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: non-inferiority double-blinded, randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPO Tri Fluvac vaccine (Active Comparator): 408 participants will receive a seasonal trivalent inactivated split virion influenza vaccine recommended for Southern Hemisphere in 2020 (consisting of A/Brisbane/02/2018 (H1N1)pdm-09-like virus, A/South Australia/34/2019 (H3N2)-like virus, and B/Washington/02/2019-like (B/Victoria lineage) virus) produced by the Government Pharmaceutical Organization (GPO), Thailand. The vaccine to be administered by intramuscular (IM) injection.
  Interventions: Biological: GPO Tri Fluvac vaccine
- Licensed Influenza vaccine (Active Comparator): 408 will receive a Licensed Influenza vaccine (seasonal trivalent inactivated split virion influenza vaccine recommended for Southern Hemisphere in 2020 (consisting of A/Brisbane/02/2018 (H1N1) pdm-09-like virus, A/South Australia/34/2019 (H3N2)-like virus, and B/Washington/02/2019-like (B/Victoria lineage) virus) 0.5 mL administered intramuscularly (IM) in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Licensed influenza vaccine

INTERVENTIONS:
Biological: GPO Tri Fluvac vaccine — Each dose of Tri Fluvac contains a total of 45 micrograms (μg) hemagglutinin (HA) per 0.5 ml dose (15 μg HA per strain per dose), to be administered by intramuscular (IM) injection. Tri Fluvac is manufactured and formulated into a multiple-dose vial vaccine (2 doses) using thimerosal at relatively low concentration as preservative (≤ 5.75 μg mercury/ dose). Each 0.5 ml dose of vaccine may contain residual amounts of ovalbumin (≤ 1.0μg), formaldehyde (≤ 100μg), tween 80 (≤ 0.9μg), triton x-100 (≤0.05μg) and gentamicin (≤0.075μg).
  Arms: GPO Tri Fluvac vaccine
Biological: Licensed influenza vaccine — The comparator licensed influenza vaccine is a seasonal trivalent inactivated split virion influenza vaccine recommended for Southern Hemisphere in 2020
  Arms: Licensed Influenza vaccine

SUMMARY:
The study is aim to evaluate the Immunogenicity with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza vaccine).

DETAILED DESCRIPTION:
This is a phase III, non-inferiority double-blinded, randomized, controlled trial of immunogenicity with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza vaccine).

A total of about 816 healthy Thai male and female adult volunteers ≥ 65 years of age; 408 participants will be randomized to receive the GPO Tri Fluvac and 408 will receive an active comparator (a 1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old on the day of screening, having Thai ID card or equivalent
* Able to read and write in Thai and sign written informed consent form
* Able to attend all scheduled visits and to comply with all trial procedures.
* Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable, under control or unchanged for the past three months. If medication is used to treat the condition, the medication dose must have been stable for at least one month preceding vaccination.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Hypersensitivity after previous administration of any vaccine.
* Having a history of H1N1, H3N2 or FluB infection within 3 months preceding enrollment to the trial
* Vaccination against influenza in the past 6 months preceding enrollment to the trial
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 28 visit.
* History of bronchial asthma, chronic lung diseases, chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression < 6 months prior to immunization
* History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. egg proteins, gentamicin or thimerosal)
* History of Guillain-Barré Syndrome or cerebrovascular events
* Having acute infection with fever > 38 degree Celsius or noninfectious diseases (within 72 hours) preceding enrollment in the trial
* Volunteers who have been taking immunoglobulin products or have had a blood transfusion during past 3 months before the beginning of the trial or planned receipt of such products prior to the Day 28 visit.
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine
* Study site employees who are involved in the protocol and/or may have direct access to study related area

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of seroconverted participants at 28 days post vaccination | 28 days
  seroconversion is defined as a serum HI antibody titer meeting the following four fold rising criteria:
  * Pre-vaccination titer <1:10 and a post-vaccination measured on Day 28 of ≥1:40; or
  * Pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination measured on Day 28.
Geometric Mean Titers (GMTs) of serum HI antibodies at baseline (Day 0) and post- vaccination (Day 28). | 28 days
  Geometric mean titers (GMTs) of serum HI antibodies pre- (Day 0) and post-vaccination (Day 28) for each of the three vaccine antigens. GMTs will be calculated with 95% CI.

SECONDARY OUTCOMES:
Number and percentage of participants with solicited local and systemic adverse events. post vaccination | 30 minutes, Day 1-3 post-vaccination
  Solicited local adverse events including redness/erythema, swelling/induration, pain, and limitation of arm movement. Solicited systemic adverse events including fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, and headache.
Number and percentage of participants with unsolicited adverse event. | 180 days
  Number and percentage of participants with unsolicited adverse event occuring during the entire study period (Days 0-180)
Number and percentage of participants with serious adverse event. | 180 days
  Number and percentage of participants with serious adverse event occuring during the entire study period (Days 0-180)
Number and percentage of participants with HI response with and without pre-existing HI antibody. | 28 days
  Number and percentage of participants with a HI antibody titer ≥1:40 (seroprotective level) to each of the three vaccine antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Principal Investigator — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University,
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No